CLINICAL TRIAL: NCT00968526
Title: Safety and Immunogenicity Study of GSK Biologicals' Influenza Vaccine GSK2340272A in Adults Aged 18 Years and Above
Brief Title: Study to Evaluate Immunogenicity and Safety of an Investigational Influenza Vaccine (H1N1) in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113459; 2009-013837-92 (EudraCT Number)
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Influenza
Keywords: influenza infection; GSK Bio's influenza vaccine GSK2340272A
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- GSK2340272A 2D Group (Experimental): Healthy male or female adults, aged 18 to 60 years (18-60y) and above (>60y), who received two doses (2D) of GSK2340272A vaccine, one administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and the other one, administered intramuscularly in the deltoid region of the dominant arm at Day 21.
  Interventions: Biological: GSK investigational vaccine GSK2340272A
- GSK2340272A 1D Group (Experimental): Healthy male or female adults, aged 18 to 60 years (18-60y) and above (>60y), who received a single dose (1D) of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0.
  Interventions: Biological: GSK investigational vaccine GSK2340272A

INTERVENTIONS:
Biological: GSK investigational vaccine GSK2340272A — One or two intramuscular injections in the deltoid region of the non-dominant or the dominant arm.

SUMMARY:
The objective of the study is to evaluate the immunogenicity and safety of GSK Biologicals' investigational vaccine GSK2340272A.

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged 18 years or above at the time of the first vaccination.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Satisfactory baseline medical assessment by history and physical examination. Stable health status is defined as the absence of a health event satisfying the definition of a serious adverse event, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within one month prior to enrolment.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period. Potential subjects in the follow-up phase of a prior investigational study may be enrolled if the investigator's judgment is that it will have no effect on safety, reactogenicity, or immunogenicity endpoints in this study, and that it does not violate the protocol requirements of the prior trial.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an axillary temperature >= 37.5ºC, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination. NOTE: The subject may be vaccinated at a later date, provided symptoms have resolved, vaccination occurs within the window specified by the protocol, and all other eligibility criteria continue to be satisfied.
* Diagnosed with cancer, or treatment for cancer, within the past 3 years.
* Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
* Persons with a history of histological-confirmed basal cell carcinoma of the skin successfully treated with local excision only are excepted and may enrol within 3 years of diagnosis, but other histological types of skin cancer require a 3-year untreated and disease-free window as above.
* Women who are disease-free 3 years or more after treatment for breast cancer and receiving long-term prophylactic hormonal therapy are excepted and may enrol.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Chronic administration of immunosuppressants or other immune modifying drugs within 6 months of study enrolment or planned administration during the study period.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrolment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome.
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start.
* Administration of any vaccines within 30 days before vaccination.
* Any known or suspected allergy to any constituent of influenza vaccines; anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-09-08 (Actual); Primary Completion 2010-09-23 (Actual); Study Completion 2010-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Van Damme P, Kafeja F, Bambure V, Hanon E, Moris P, Roman F, Gillard P. Long-term persistence of humoral and cellular immune responses induced by an AS03A-adjuvanted H1N1 2009 influenza vaccine: an open-label, randomized study in adults aged 18-60 years and older. Hum Vaccin Immunother. 2013 Jul;9(7):1512-22. doi: 10.4161/hv.24504. Epub 2013 Apr 9. PMID 23571166
- [Background] Roman F, Vaman T, Kafeja F, Hanon E, Van Damme P. AS03(A)-Adjuvanted influenza A (H1N1) 2009 vaccine for adults up to 85 years of age. Clin Infect Dis. 2010 Sep 15;51(6):668-77. doi: 10.1086/655830. PMID 20687838
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 113459 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113459 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113459 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113459 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113459 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113459 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113459 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At Day 21, all subjects had received 1 dose of GSK2340272A vaccine and therefore no distinction was made between groups for the Day 21 analysis.
Period: Overall Study
Arm/Group | GSK2340272A 2D Group | GSK2340272A 1D Group
Started | 138 | 102
Completed | 135 | 102
Not Completed | 3 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Migrated/moved from study area | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340272A 2D Group | GSK2340272A 1D Group | Total
Number analyzed (Participants) | 138 | 102 | 240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.0 (18.2) | 53.6 (18.3) | 54.4 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 49 | 117
  Male | 70 | 53 | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Caucasian/European heritage | 138 | 102 | 240

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted (SCR) Subjects for Hemagglutination Inhibition (HI) Antibodies
Description: Seroconversion was defined as: For initially seronegative subjects [antibody titer (below) < 10 post-vaccination], antibody titer greater than or equal to (≥) 40 after vaccination; For initially seropositive subjects (antibody titer ≥ 10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09). This outcome included only subjects who received two doses of the study product and results were tabulated per age stratum. The CHMP criterion was fulfilled if the post-vaccination point estimate for SPR was > 70% in subjects 18 to 60 of age or > 60% for subjects above 60 years of age .
Time Frame: At Day 21
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 42, which included all evaluable subjects for whom 2 doses were administrated and the assay results were available for antibodies against H1N1 antigen for blood sample taken 21 or 42 days after the first vaccine dose and 21 days after the second dose.
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340272A 2D (18-60y) Sub-Group: Sub-Group of healthy male or female adults, aged 18 to 60 years (18-60y), who received two doses (2D) of GSK2340272A vaccine, one administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and the other one, administered intramuscularly in the deltoid region of the dominant arm at Day 21.
- GSK2340272A 2D (>60y) Sub-Group: Sub-Group of healthy male or female adults, above 60 years (>60y), who received two doses 2D of GSK2340272A vaccine, one administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and the other one, administered intramuscularly in the deltoid region of the dominant arm at Day 21.
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group
Number analyzed (Participants) | 66 | 67
Participants | 63 | 53

2. Primary Outcome: Number of Subjects Who Were Seroprotected (SPR) for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40, that usually is accepted as indicating protection. This outcome included only subjects who received two doses of the study product and the results were tabulated per age stratum. The CHMP criterion was fulfilled if the post-vaccination point estimate for SPR was > 70% in subjects 18 to 60 of age or > 60% for subjects above 60 years of age .
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom 2 doses were administrated and the assay results were available for antibodies against H1N1 antigen for blood sample taken 21 or 42 days after the first vaccine dose and 21 days after the second vaccine dose.
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340272A 2D (>60y) Sub-Group: Sub-Group of healthy male or female adults, above 60 years (>60y), who received two doses (2D) of GSK2340272A vaccine, one administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and the other one, administered intramuscularly in the deltoid region of the dominant arm at Dat 21.
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group
Number analyzed (Participants) | 66 | 67
Participants | 65 | 59

3. Primary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: GMFR was defined as the fold change in serum HI geometric mean titers (GMTs) post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/CAL/7/09. This outcome included only subjects who received two doses of the study product and results were tabulated per age stratum. The CHMP criterion was fulfilled if the point estimated for GMFR was > 2.5 in subjects 18 to 60 years old or > 2 for subjects > 60 years of age.
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Groups:
- GSK2340272A 2D (>60y) Sub-Group: Sub-Group of healthy male or female adults, above 60 years (>60y), who received two doses (2D) of GSK2340272A vaccine, one administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and the other one, administered intramuscularly in the deltoid region of the dominant arm at Day 21.
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group
Number analyzed (Participants) | 66 | 67
Fold change | 38.71 [29.10 to 51.51] | 13.86 [10.29 to 18.65]

4. Secondary Outcome: Number of Subjects Who Were Seropositive for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seropositive subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:10, that usually is accepted as indicating protection. The results for this assay were tabulated per age stratum.
Time Frame: At Days 0, 21 and 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom 1 dose and 2 doses were administered and the assay results were available for antibodies against H1N1 antigen for blood sample taken 21 or 42 days after the first vaccine dose and 21 days after the second vaccine dose.
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340272A 1D (18-60y) Sub-Group: Sub-Group of healthy male or female adults, aged 18 to 60 years (18-60y), who received a single dose (1D) of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0.
- GSK2340272A 1D (>60y) Sub-Group: Sub-Group of healthy male or female adults, aged above 60 years (>60y), who received a single dose (1D) of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0.
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 66 | 67 | 50 | 49
Participants
  Flu A/California/7/2009, Day 0 | 24 | 28 | 20 | 21
  Flu A/California/7/2009, Day 21 | 66 | 67 | 50 | 47
  Flu A/California/7/2009, Day 42 | 66 | 67 | 50 | 48

5. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/CAL/7/09. The reference seropositivity cut-off value was ≥ 1:10. The results for this assay were tabulated per age stratum.
Time Frame: At Days 0, 21 and 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom 1 dose and 2 doses were administrated and the assay results were available for antibodies against H1N1 antigen for blood sample taken 21 or 42 days after the first vaccine dose and 21 days after the second vaccine dose.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- GSK2340272A 1D (>60y) Sub-Group: Sub-Group of healthy male or female adults, above 60 years (>60y), who received a single dose (1D) of GSK2340272A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm at Day 0.
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 66 | 67 | 50 | 49
Titers
  Flu A/CAL/7/09, Day 0 | 8.8 [7.0 to 10.9] | 10.3 [7.7 to 13.7] | 8.6 [6.8 to 10.8] | 9.7 [7.3 to 13.0]
  Flu A/CAL/7/09, Day 21 | 339.1 [258.6 to 444.8] | 142.7 [108.5 to 187.8] | 388.6 [262.0 to 576.2] | 129.3 [89.9 to 186.0]
  Flu A/CAL/7/09, Day 42 | 610.6 [507.9 to 734.0] | 345.8 [278.0 to 430.1] | 331.2 [220.7 to 497.1] | 117.1 [82.4 to 166.4]

6. Secondary Outcome: Number of Subjects Who Were Seropositive for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: as for outcome 4
Time Frame: At Day 182 and 364
Population: The analysis was performed on the ATP cohort for persistence at Day 182 and 364, which included all evaluable subjects for whom data concerning immunogenicity outcome measure and assay results for antibodies against the study vaccine antigen component at Day 182 and 364 were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 67 | 68 | 52 | 50
Participants
  Flu A/California/7/2009, Day 182: number analyzed (Participants) | 67 | 68 | 51 | 50
  Flu A/California/7/2009, Day 182 | 67 | 68 | 51 | 46
  Flu A/California/7/2009, Day 364 | 67 | 65 | 44 | 41

7. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: as for outcome 5
Time Frame: At Day 182 and 364
Population: The analysis was performed on the ATP cohort for persistence at Day 182 and 364, which included all evaluable subjects for whom data concerning immunogenicity outcome measure and whom assay results for antibodies against the study vaccine antigen component at Day 182 and 364 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 67 | 68 | 52 | 50
Titers
  Flu A/CAL/7/09, Day 182: number analyzed (Participants) | 67 | 68 | 51 | 50
  Flu A/CAL/7/09, Day 182 | 214.8 [169.8 to 271.8] | 108.7 [85.7 to 137.8] | 143.5 [96.6 to 213.0] | 51.6 [34.9 to 76.5]
  Flu A/CAL/7/09, Day 364 | 90.5 [69.4 to 118.1] | 42.3 [32.6 to 54.8] | 64.2 [41.3 to 99.7] | 28.1 [19.4 to 40.6]

8. Secondary Outcome: Number of Seroconverted (SCR) Subjects for Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/2009 Strain of Influenza Disease
Description: Seroconversion was defined as: For initially seronegative subjects [antibody titer below (<) 10 post to vaccination], antibody titer greater than or equal to (≥) 40 after vaccination; For initially seropositive subjects (antibody titer ≥ 10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09). This outcome included only subjects who received one dose of the study product and the results were tabulated per age stratum. The CHMP criterion was fulfilled if the post-vaccination point estimate for SPR was > 70% in subjects 18 to 60 of age or > 60% for subjects above 60 years of age .
Time Frame: At Days 21 and 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom 1 dose was administrated and the assay results were available for antibodies against H1N1 antigen for blood sample taken 21 days and 42 days after the first vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 50 | 49
Participants
  Flu A/CAL/7/2009, Day 21 | 47 | 38
  Flu A/CAL/7/2009, Day 42 | 46 | 39

9. Secondary Outcome: Number of Seroconverted (SCR) Subjects for Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: Seroconversion was defined as: For initially seronegative subjects [antibody titer below (<) 10 post to vaccination], antibody titer greater than or equal to (≥) 40 after vaccination; For initially seropositive subjects (antibody titer ≥ 10 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was A/California/7/2009 (H1N1)v-like influenza (Flu A/CAL/7/09). The results for this assay were tabulated per age stratum. The CHMP criterion was fulfilled if the post-vaccination point estimate for SPR was > 70% in subjects 18 to 60 of age or > 60% for subjects above 60 years of age .
Time Frame: At Days 182 and 364
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 67 | 68 | 52 | 50
Participants
  Flu A/CAL/7/09, Day 182: number analyzed (Participants) | 67 | 68 | 51 | 50
  Flu A/CAL/7/09, Day 182 | 63 | 52 | 42 | 21
  Flu A/CAL/7/09, Day 364 | 50 | 28 | 32 | 15

10. Secondary Outcome: Number of Subjects Who Were Seroprotected (SPR ) for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40, that usually is accepted as indicating protection. This outcome included only subjects who received one dose of the study product and the results were tabulated per age stratum. The CHMP criterion was fulfilled if the post-vaccination point estimate for SPR was > 70% in subjects 18 to 60 of age or > 60% for subjects above 60 years of age .
Time Frame: At Days 0, 21 and 42
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom 1 dose was administrated and the assay results were available for antibodies against H1N1 antigen for blood sample taken 21 and 42 days after the first vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 50 | 49
Participants
  Flu A/California/7/2009, Day 0 | 4 | 5
  Flu A/California/7/2009, Day 21 | 48 | 42
  Flu A/California/7/2009, Day 42 | 47 | 43

11. Secondary Outcome: Number of Subjects Who Were Seroprotected (SPR ) for HI Antibodies Against the Flu A/California/7/2009 (H1N1) Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40, that usually is accepted as indicating protection. The results for this assay were tabulated per age stratum. The CHMP criterion was fulfilled if the post-vaccination point estimate for SPR was > 70% in subjects 18 to 60 of age or > 60% for subjects above 60 years of age.
Time Frame: At Days 182 and 364
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 67 | 68 | 52 | 50
Participants
  Flu A/California/7/2009, Day 182: number analyzed (Participants) | 67 | 68 | 51 | 50
  Flu A/California/7/2009, Day 182 | 65 | 61 | 44 | 28
  Flu A/California/7/2009, Day 364 | 53 | 37 | 34 | 22

12. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: GMFR was defined as the fold change in serum HI geometric mean titers (GMTs) post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/CAL/7/09. This outcome included only subjects who received one dose of the study product and the results were tabulated per age stratum. The CHMP criterion was fulfilled if the point estimated for GMFR was > 2.5 in subjects 18 to 60 years old or > 2 for subjects > 60 years of age.
Time Frame: At Days 21 and 42
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 50 | 49
Fold change
  Flu A/CAL/7/09, Day 21 | 45.30 [30.32 to 67.68] | 13.32 [9.04 to 19.61]
  Flu A/CAL/7/09, Day 42 | 38.62 [25.96 to 57.45] | 12.06 [8.39 to 17.33]

13. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against Flu A/CAL/7/09 Strain of Influenza Disease
Description: GMFR was defined as the fold change in serum HI geometric mean titers (GMTs) post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/CAL/7/09. The results for this assay were tabulated per age stratum. The CHMP criterion was fulfilled if the point estimated for GMFR was > 2.5 in subjects 18 to 60 years old or > 2 for subjects > 60 years of age.
Time Frame: At Day 182 and 364
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 67 | 68 | 52 | 50
Fold change
  Flu A/CAL/7/09, Day 182: number analyzed (Participants) | 67 | 68 | 51 | 50
  Flu A/CAL/7/09, Day 182 | 24.73 [19.31 to 31.67] | 10.45 [8.24 to 13.24] | 17.14 [11.83 to 24.84] | 5.31 [3.73 to 7.56]
  Flu A/CAL/7/09, Day 364 | 10.4 [8.1 to 13.4] | 4.3 [3.5 to 5.2] | 7.6 [5.1 to 11.5] | 2.9 [2.1 to 4.0]

14. Secondary Outcome: Number of Seropositive Subjects for Serum Neutralizing Antibodies Against Flu A/Netherlands (Neth)/602/09
Description: A seropositive subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:8, that usually is accepted as indicating protection. The Flu strain assessed was Flu A/Neth/602/09. The results for this assay were tabulated per age stratum.
Time Frame: At Days 0, 21, 42 and 182
Population: The analysis was performed on the ATP cohort for persistence at Day 182, which included all evaluable subjects for whom data concerning immunogenicity outcome measure and assay results for antibodies against the study vaccine antigen component at Day 182 were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 22 | 22 | 17 | 18
Participants
  Flu A/Neth/602/09, Day 0 | 16 | 17 | 11 | 12
  Flu A/Neth/602/09, Day 21 | 21 | 22 | 17 | 18
  Flu A/Neth/602/09, Day 42 | 22 | 22 | 17 | 18
  Flu A/Neth/602/09, Day 182 | 21 | 22 | 16 | 16

15. Secondary Outcome: Titers for Serum Neutralizing Antibodies Against Flu A/Neth/602/09 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The flu strain assessed was Flu A/Neth/602/09. The reference seropositivity cut-off value was ≥ 1:8. The results for this assay were tabulated per age stratum.
Time Frame: At Days 0, 21, 42 and 182
Population: The analysis was performed on the ATP cohort for persistence at Day 182, which included all evaluable subjects for whom data concerning immunogenicity outcome measures and assay results for antibodies against the study vaccine antigen component at Day 182 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 22 | 22 | 17 | 18
Titers
  Flu A/Neth/602/09, Day 0 | 11.9 [8.0 to 17.8] | 16.9 [10.1 to 28.1] | 12.6 [6.7 to 23.9] | 21.3 [10.1 to 44.9]
  Flu A/Neth/602/09, Day 21 | 199.8 [94.1 to 424.2] | 169.7 [85.6 to 336.5] | 199.1 [92.3 to 429.7] | 83.5 [38.8 to 179.4]
  Flu A/Neth/602/09, Day 42 | 326.8 [183.0 to 583.3] | 309.5 [189.3 to 505.9] | 136.7 [64.8 to 288.6] | 86.7 [48.0 to 156.7]
  Flu A/Neth/602/09, Day 182 | 128.7 [73.5 to 225.2] | 96.7 [59.3 to 157.5] | 55.2 [24.7 to 123.3] | 65.3 [30.8 to 138.4]

16. Secondary Outcome: Number of Seroconverted Subjects for Serum Neutralizing Antibodies Against Flu A/Neth/602/09
Description: Seroconversion was defined as: For initially seronegative subjects, antibody titer ≥ 1:8 after vaccination; For initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer. The Flu strain assessed was Flu A/Neth/602/09. The results were tabulated per age stratum.
Time Frame: At Days 21, 42 and 182
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 22 | 22 | 17 | 18
Participants
  Flu A/Neth/602/09, Day 21 | 15 | 15 | 12 | 6
  Flu A/Neth/602/09, Day 42 | 20 | 19 | 11 | 5
  Flu A/Neth/602/09, Day 182 | 18 | 14 | 6 | 7

17. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. This outcome included all the subjects who received 1 dose of the study product and the assay results were tabulated per age stratum.
Time Frame: During the 7-day (Days 0-6) post-dose 1 vaccination period
Population: The analysis was performed on the Total Vaccinated cohort (TVc), which included all vaccinated subjects who filled in their symptom sheets. The results were tabulated for the pooled groups and per age stratum, because until Day 21 no distinction was made in terms of study groups, since all subjects had received 1 dose of GSK2340272A vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340272A 1D & 2D (18-60y) Sub-Group: Pooled group for healthy male or female adults, aged 18 to 60 years (18-60y), who received a single dose (1D) or two doses (2D) of GSK2340272A vaccine, one administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and the other one, administered intramuscularly in the deltoid region of the dominant arm at Day 21.
- GSK2340272A 1D & 2D (>60y) Sub-Group: Pooled group for healthy male or female adults, above 60 years (>60y), who received a single dose 1D or two doses 2D of GSK2340272A vaccine, one administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and the other one, administered intramuscularly in the deltoid region of the dominant arm at Day 21.
Arm/Group | GSK2340272A 1D & 2D (18-60y) Sub-Group | GSK2340272A 1D & 2D (>60y) Sub-Group
Number analyzed (Participants) | 120 | 120
Participants
  Any Pain | 105 | 78
  Grade 3 Pain | 0 | 0
  Any Redness | 1 | 9
  Grade 3 Redness | 0 | 0
  Any Swelling | 11 | 12
  Grade 3 Swelling | 0 | 0

18. Secondary Outcome: Number of Days With Solicited Local Symptoms
Description: The number of days with any solicited local symptoms reported during the solicited post-vaccination period. This outcome included all the subjects who received 1 dose of the study product and the assay results were tabulated per age stratum.
Time Frame: During the 7-day (Days 0-6) post-dose 1 vaccination period
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK2340272A 1D & 2D (18-60y) Sub-Group | GSK2340272A 1D & 2D (>60y) Sub-Group
Number analyzed (Participants) | 105 | 82
Days
  Pain: number analyzed (Participants) | 105 | 78
  Pain | 3.0 [2.0 to 4.0] | 2.5 [1.0 to 4.0]
  Redness: number analyzed (Participants) | 1 | 9
  Redness | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 3.0]
  Swelling: number analyzed (Participants) | 11 | 12
  Swelling | 2.0 [2.0 to 2.0] | 2.0 [1.0 to 2.0]

19. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. This outcome included only subjects who received two doses of the study product and the results were tabulated per age stratum.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on a subset of subjects from the Total Vaccinated cohort (TVc), which included all subjects who received 2 doses of GSK2340272A vaccine and who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group
Number analyzed (Participants) | 68 | 70
Participants
  Any Pain, Dose 1 | 57 | 46
  Grade 3 Pain, Dose 1 | 0 | 0
  Any Redness, Dose 1 | 0 | 3
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 5 | 4
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2 | 51 | 42
  Grade 3 Pain, Dose 2 | 2 | 0
  Any Redness, Dose 2 | 1 | 5
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2 | 3 | 3
  Grade 3 Swelling, Dose 2 | 0 | 1
  Any Pain, Across doses | 61 | 52
  Grade 3 Pain, Across doses | 2 | 0
  Any Redness, Across doses | 1 | 6
  Grade 3 Redness, Across doses | 0 | 0
  Any Swelling, Across doses | 7 | 6
  Grade 3 Swelling, Across doses | 0 | 1

20. Secondary Outcome: Number of Days With Solicited Local Symptoms
Description: The number of days with any solicited local symptoms reported during the solicited post-vaccination period. This outcome included only subjects who received 2 doses of the study product and the results were tabulated per age stratum. No subjects from GSK2340272A 2D (18-60y) Sub-Group presented any redness post dose 1.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on a subset of subjects from the Total Vaccinated cohort (TVc), which included all subjects who received 2 doses of GSK2340272A and who filled in their symptom sheets.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group
Number analyzed (Participants) | 68 | 70
Days
  Pain, Dose 1 | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 3.0]
  Pain, Dose 2 | 3.0 [2.0 to 3.0] | 2.0 [1.0 to 3.0]
  Pain, Overall/dose | 3.0 [2.0 to 3.5] | 2.0 [1.0 to 3.0]
  Redness, Dose 1 | 0 [0 to 0] | 1.0 [1.0 to 3.0]
  Redness, Dose 2 | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 2.0]
  Redness, Overall/dose | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.5]
  Swelling, Dose 1 | 2.0 [2.0 to 2.0] | 2.0 [1.5 to 2.5]
  Swelling, Dose 2 | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 1.0]
  Swelling, Overall/dose | 2.0 [1.5 to 2.5] | 1.0 [1.0 to 2.0]

21. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating and fever [defined as axillary temperature equal to or above (>) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = temperature ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination. This outcome included all the subjects who received 1 dose of the study product and the assay results were tabulated per age stratum.
Time Frame: During the 7-day (Days 0-6) post-dose 1 vaccination period
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 1D & 2D (18-60y) Sub-Group | GSK2340272A 1D & 2D (>60y) Sub-Group
Number analyzed (Participants) | 120 | 120
Participants
  Any Fatigue | 43 | 26
  Grade 3 Fatigue | 2 | 1
  Related Fatigue | 40 | 24
  Any Headache | 44 | 22
  Grade 3 Headache | 1 | 0
  Related Headache | 43 | 21
  Any Joint pain | 19 | 17
  Grade 3 Joint pain | 0 | 1
  Related Joint pain | 17 | 14
  Any Muscle aches | 29 | 25
  Grade 3 Muscle aches | 2 | 1
  Related Muscle aches | 25 | 23
  Any Shivering | 23 | 7
  Grade 3 Shivering | 0 | 0
  Related Shivering | 22 | 7
  Any Sweating | 19 | 6
  Grade 3 Sweating | 1 | 0
  Related Sweating | 17 | 6
  Any Temperature | 1 | 0
  Grade 3 Temperature | 0 | 0
  Related Temperature | 1 | 0

22. Secondary Outcome: Number of Days With Solicited General Symptoms
Description: The number of days with any solicited general symptoms reported during the solicited post-vaccination period. This outcome included all the subjects who received 1 dose of the study product and the results were tabulated per age stratum.
Time Frame: During the 7-day (Days 0-6) post-dose 1 vaccination period
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK2340272A 1D & 2D (18-60y) Sub-Group | GSK2340272A 1D & 2D (>60y) Sub-Group
Number analyzed (Participants) | 78 | 52
Days
  Fatigue: number analyzed (Participants) | 43 | 26
  Fatigue | 2.0 [1.0 to 4.0] | 1.5 [1.0 to 2.0]
  Headache: number analyzed (Participants) | 44 | 22
  Headache | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Joint pain: number analyzed (Participants) | 19 | 17
  Joint pain | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0]
  Muscle aches: number analyzed (Participants) | 29 | 25
  Muscle aches | 2.0 [2.0 to 4.0] | 3.0 [1.0 to 4.0]
  Shivering: number analyzed (Participants) | 23 | 7
  Shivering | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]
  Sweating: number analyzed (Participants) | 19 | 6
  Sweating | 2.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0]
  Temperature: number analyzed (Participants) | 6 | 1
  Temperature | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0]

23. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating and fever [defined as axillary temperature above (>) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = temperature ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination. This outcome inlcuded only subjects who received two doses of the study product and the results were tabulated per age stratum.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group
Number analyzed (Participants) | 68 | 70
Participants
  Any Fatigue, Dose 1 | 24 | 15
  Grade 3 Fatigue, Dose 1 | 2 | 0
  Related Fatigue, Dose 1 | 21 | 14
  Any Headache, Dose 1 | 23 | 12
  Grade 3 Headache, Dose 1 | 1 | 0
  Related Headache, Dose 1 | 22 | 11
  Any Joint pain, Dose 1 | 12 | 9
  Grade 3 Joint pain, Dose 1 | 0 | 0
  Related Joint pain, Dose 1 | 10 | 6
  Any Muscle aches, Dose 1 | 19 | 12
  Grade 3 Muscle aches, Dose 1 | 1 | 0
  Related Muscle aches, Dose 1 | 15 | 10
  Any Shivering, Dose 1 | 14 | 2
  Grade 3 Shivering, Dose 1 | 0 | 0
  Related Shivering, Dose 1 | 13 | 2
  Any Sweating, Dose 1 | 12 | 5
  Grade 3 Sweating, Dose 1 | 1 | 0
  Related Sweating, Dose 1 | 11 | 5
  Any Temperature, Dose 1 | 1 | 0
  Grade 3 Temperature, Dose 1 | 0 | 0
  Related Temperature, Dose 1 | 1 | 0
  Any Fatigue, Dose 2 | 19 | 15
  Grade 3 Fatigue, Dose 2 | 2 | 0
  Related Fatigue, Dose 2 | 19 | 15
  Any Headache, Dose 2 | 15 | 12
  Grade 3 Headache, Dose 2 | 1 | 0
  Related Headache, Dose 2 | 15 | 12
  Any Joint pain, Dose 2 | 11 | 13
  Grade 3 Joint pain, Dose 2 | 1 | 0
  Related Joint pain, Dose 2 | 11 | 13
  Any Muscle aches, Dose 2 | 15 | 13
  Grade 3 Muscle aches, Dose 2 | 1 | 0
  Related Muscle aches, Dose 2 | 15 | 13
  Any Shivering, Dose 2 | 18 | 5
  Grade 3 Shivering, Dose 2 | 2 | 1
  Related Shivering, Dose 2 | 18 | 5
  Any Sweating, Dose 2 | 11 | 5
  Grade 3 Sweating, Dose 2 | 1 | 0
  Related Sweating, Dose 2 | 11 | 5
  Any Temperature, Dose 2 | 2 | 0
  Grade 3 Temperature, Dose 2 | 0 | 0
  Related Temperature, Dose 2 | 2 | 0
  Any Fatigue, Across doses | 29 | 26
  Grade 3 Fatigue, Across doses | 3 | 0
  Related Fatigue, Across doses | 27 | 25
  Any Headache, Across doses | 29 | 20
  Grade 3 Headache, Across doses | 2 | 0
  Related Headache, Across doses | 28 | 19
  Any Joint pain, Across doses | 16 | 18
  Grade 3 Joint pain, Across doses | 1 | 0
  Related Joint pain, Across doses | 15 | 16
  Any Muscle aches, Across doses | 26 | 22
  Grade 3 Muscle aches, Across doses | 2 | 0
  Related Muscle aches, Across doses | 23 | 20
  Any Shivering, Across doses | 22 | 7
  Grade 3 Shivering, Across doses | 2 | 1
  Related Shivering, Across doses | 21 | 7
  Any Sweating, Across doses | 19 | 9
  Grade 3 Sweating, Across doses | 2 | 0
  Related Sweating, Across doses | 18 | 9
  Any Temperature, Across doses | 3 | 0
  Grade 3 Temperature, Across doses | 0 | 0
  Related Temperature, Across doses | 3 | 0

24. Secondary Outcome: Number of Days With Solicited General Symptoms
Description: The number of days with any solicited general symptoms reported during the solicited post-vaccination period. This outcome included only subjects who received two doses of the study product and the results were tabulated per age stratum. No subjects from GSK2340272A 2D (>60y) Sub-Group reported any temperature.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 19
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group
Number analyzed (Participants) | 68 | 70
Days
  Fatigue, Dose 1 | 2.0 [1.5 to 4.5] | 1.0 [1.0 to 2.0]
  Fatigue, Dose 2 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Fatigue, Overall/dose | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 2.0]
  Headache, Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.5]
  Headache, Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Headache, Overall/dose | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0]
  Joint pain, Dose 1 | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 5.0]
  Joint pain, Dose 2 | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Joint pain, Overall/dose | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Muscle aches, Dose 1 | 2.0 [2.0 to 4.0] | 2.5 [1.0 to 4.5]
  Muscle aches, Dose 2 | 2.0 [2.0 to 3.0] | 1.0 [1.0 to 3.0]
  Muscle aches, Overall/dose | 2.0 [2.0 to 4.0] | 1.0 [1.0 to 4.0]
  Sweating, Dose 1 | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Sweating, Dose 2 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0]
  Sweating, Overall/dose | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Shivering, Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Shivering, Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Shivering, Overall/dose | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Temperature, Dose 1 | 1.0 [1.0 to 1.0] | NA [NA to NA] — No subjects from GSK2340272A (>60y) Sub-Group reported any temperature for dose 1.
  Temperature, Dose 2 | 2.0 [2.0 to 2.0] | NA [NA to NA] — No subjects from GSK2340272A (>60y) Sub-Group reported any temperature for dose 2.
  Temperature, Overall/dose | 2.0 [1.0 to 2.0] | NA [NA to NA] — No subjects from GSK2340272A (>60y) Sub-Group reported any temperature across doses.

25. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESIs)
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration. The results were tabulated per age stratum.
Time Frame: During the entire study period (from Day 0 up to Day 364)
Population: The analysis was performed on the Total Vaccinated cohort (TVc), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 68 | 70 | 52 | 50
Participants | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Subjects With Normal/Abnormal Biochemical and Haematological Levels
Description: Among biochemical and haematological parameters assessed were alanine aminotransferase [ALT], alkaline phosphatase [AP], aspartate aminotransferase [AST], total bilirubin [BIL], creatinine [CRE], blood urea nitrogen [BUN]. Levels of haematological/biochemical parameters assessed with respect to normal laboratory values were - unknown, below, within and above in subjects aged 18-60 years and > 60 years old.
Time Frame: At Days 0, 21, 42, 182 and 364
Population: The analysis was performed on the Total Vaccinated cohort (TVc), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 68 | 70 | 52 | 50
Participants
  ALT, Day 0: Unknown | 0 | 0 | 0 | 0
  ALT, Day 0: Below | 0 | 0 | 0 | 0
  ALT, Day 0: Within | 56 | 66 | 44 | 48
  ALT, Day 0: Above | 12 | 4 | 8 | 2
  ALT, Day 21: Unknown | 0 | 0 | 0 | 0
  ALT, Day 21: Below | 0 | 0 | 0 | 0
  ALT, Day 21: Within | 56 | 65 | 45 | 46
  ALT, Day 21: Above | 12 | 5 | 7 | 4
  ALT, Day 42: Unknown | 0 | 0 | 0 | 0
  ALT, Day 42: Below | 0 | 0 | 0 | 0
  ALT, Day 42: Within | 57 | 68 | 46 | 44
  ALT, Day 42: Above | 11 | 2 | 6 | 6
  ALT, Day 182: number analyzed (Participants) | 67 | 69 | 52 | 50
  ALT, Day 182: Unknown | 0 | 0 | 0 | 0
  ALT, Day 182: Below | 0 | 0 | 0 | 0
  ALT, Day 182: Within | 57 | 63 | 47 | 48
  ALT, Day 182: Above | 10 | 6 | 5 | 2
  ALT, Day 364: number analyzed (Participants) | 67 | 68 | 52 | 50
  ALT, Day 364: Unknown | 0 | 0 | 0 | 0
  ALT, Day 364: Below | 0 | 0 | 0 | 0
  ALT, Day 364: Within | 58 | 65 | 47 | 47
  ALT, Day 364: Above | 9 | 3 | 5 | 3
  AP, Day 0: Unknown | 0 | 0 | 0 | 0
  AP, Day 0: Below | 0 | 0 | 0 | 0
  AP, Day 0: Within | 67 | 70 | 51 | 45
  AP, Day 0: Above | 1 | 0 | 1 | 5
  AP, Day 21: Unknown | 0 | 0 | 0 | 0
  AP, Day 21: Below | 0 | 0 | 0 | 0
  AP, Day 21: Within | 67 | 69 | 52 | 46
  AP, Day 21: Above | 1 | 1 | 0 | 4
  AP, Day 42: Unknown | 0 | 0 | 0 | 0
  AP, Day 42: Below | 0 | 0 | 0 | 0
  AP, Day 42: Within | 66 | 68 | 52 | 44
  AP, Day 42: Above | 2 | 2 | 0 | 6
  AP, Day 182: number analyzed (Participants) | 67 | 69 | 52 | 50
  AP, Day 182: Unknown | 0 | 0 | 0 | 0
  AP, Day 182: Below | 0 | 0 | 0 | 0
  AP, Day 182: Within | 65 | 66 | 51 | 45
  AP, Day 182: Above | 2 | 3 | 1 | 5
  AP, Day 364: number analyzed (Participants) | 67 | 68 | 52 | 50
  AP, Day 364: Unknown | 0 | 0 | 0 | 0
  AP, Day 364: Below | 0 | 0 | 0 | 0
  AP, Day 364: Within | 63 | 67 | 51 | 47
  AP, Day 364: Above | 4 | 1 | 1 | 3
  AST, Day 0: Unknown | 0 | 0 | 0 | 0
  AST, Day 0: Below | 0 | 0 | 0 | 0
  AST, Day 0: Within | 63 | 66 | 47 | 48
  AST, Day 0: Above | 5 | 4 | 5 | 2
  AST, Day 21: Unknown | 0 | 0 | 0 | 0
  AST, Day 21: Below | 0 | 0 | 0 | 0
  AST, Day 21: Within | 67 | 67 | 49 | 48
  AST, Day 21: Above | 1 | 3 | 3 | 2
  AST, Day 42: Unknown | 0 | 0 | 0 | 0
  AST, Day 42: Below | 0 | 0 | 0 | 0
  AST, Day 42: Within | 63 | 66 | 45 | 48
  AST, Day 42: Above | 5 | 4 | 7 | 2
  AST, Day 182: number analyzed (Participants) | 67 | 69 | 52 | 50
  AST, Day 182: Unknown | 0 | 0 | 0 | 0
  AST, Day 182: Below | 0 | 0 | 0 | 0
  AST, Day 182: Within | 62 | 64 | 47 | 48
  AST, Day 182: Above | 5 | 5 | 5 | 2
  AST, Day 364: number analyzed (Participants) | 67 | 68 | 52 | 50
  AST, Day 364: Unknown | 0 | 0 | 0 | 0
  AST, Day 364: Below | 0 | 0 | 0 | 0
  AST, Day 364: Within | 63 | 65 | 49 | 48
  AST, Day 364: Above | 4 | 3 | 3 | 2
  BIL, Day 0: Unknown | 0 | 0 | 0 | 0
  BIL, Day 0: Below | 0 | 0 | 0 | 0
  BIL, Day 0: Within | 64 | 68 | 49 | 48
  BIL, Day 0: Above | 4 | 2 | 3 | 2
  BIL, Day 21: Unknown | 0 | 0 | 0 | 0
  BIL, Day 21: Below | 0 | 0 | 0 | 0
  BIL, Day 21: Within | 64 | 66 | 49 | 49
  BIL, Day 21: Above | 4 | 4 | 3 | 1
  BIL, Day 42: Unknown | 0 | 0 | 0 | 0
  BIL, Day 42: Below | 0 | 0 | 0 | 0
  BIL, Day 42: Within | 64 | 67 | 50 | 49
  BIL, Day 42: Above | 4 | 3 | 2 | 1
  BIL, Day 182: number analyzed (Participants) | 67 | 69 | 52 | 50
  BIL, Day 182: Unknown | 0 | 0 | 0 | 0
  BIL, Day 182: Below | 0 | 0 | 0 | 0
  BIL, Day 182: Within | 65 | 68 | 51 | 50
  BIL, Day 182: Above | 2 | 1 | 1 | 0
  BIL, Day 364: number analyzed (Participants) | 67 | 68 | 52 | 50
  BIL, Day 364: Unknown | 0 | 0 | 0 | 0
  BIL, Day 364: Below | 0 | 0 | 0 | 0
  BIL, Day 364: Within | 59 | 64 | 46 | 49
  BIL, Day 364: Above | 8 | 4 | 6 | 1
  CRE, Day 0: Unknown | 0 | 0 | 0 | 0
  CRE, Day 0: Below | 0 | 0 | 0 | 0
  CRE, Day 0: Within | 59 | 52 | 50 | 42
  CRE, Day 0: Above | 9 | 18 | 2 | 8
  CRE, Day 21: Unknown | 0 | 0 | 0 | 0
  CRE, Day 21: Below | 0 | 0 | 0 | 0
  CRE, Day 21: Within | 60 | 51 | 49 | 41
  CRE, Day 21: Above | 8 | 19 | 3 | 9
  CRE, Day 42: Unknown | 0 | 0 | 0 | 0
  CRE, Day 42: Below | 0 | 0 | 0 | 0
  CRE, Day 42: Within | 60 | 54 | 51 | 41
  CRE, Day 42: Above | 8 | 16 | 1 | 9
  CRE, Day 182: number analyzed (Participants) | 67 | 69 | 52 | 50
  CRE, Day 182: Unknown | 0 | 0 | 0 | 0
  CRE, Day 182: Below | 0 | 0 | 0 | 0
  CRE, Day 182: Within | 57 | 51 | 50 | 41
  CRE, Day 182: Above | 10 | 18 | 2 | 9
  CRE, Day 364: number analyzed (Participants) | 67 | 68 | 52 | 50
  CRE, Day 364: Unknown | 0 | 0 | 0 | 0
  CRE, Day 364: Below | 0 | 0 | 0 | 0
  CRE, Day 364: Within | 63 | 60 | 52 | 45
  CRE, Day 364: Above | 4 | 8 | 0 | 5
  BUN, Day 0: Unknown | 0 | 0 | 0 | 0
  BUN, Day 0: Below | 0 | 0 | 0 | 0
  BUN, Day 0: Within | 66 | 58 | 51 | 47
  BUN, Day 0: Above | 2 | 12 | 1 | 3
  BUN, Day 21: Unknown | 0 | 0 | 0 | 0
  BUN, Day 21: Below | 0 | 0 | 0 | 0
  BUN, Day 21: Within | 66 | 59 | 51 | 42
  BUN, Day 21: Above | 2 | 11 | 1 | 8
  BUN, Day 42: Unknown | 0 | 0 | 0 | 0
  BUN, Day 42: Below | 0 | 0 | 0 | 0
  BUN, Day 42: Within | 64 | 57 | 51 | 43
  BUN, Day 42: Above | 4 | 13 | 1 | 7
  BUN, Day 182: number analyzed (Participants) | 67 | 69 | 52 | 50
  BUN, Day 182: Unknown | 0 | 0 | 0 | 0
  BUN, Day 182: Below | 0 | 0 | 0 | 0
  BUN, Day 182: Within | 67 | 59 | 50 | 43
  BUN, Day 182: Above | 0 | 10 | 2 | 7
  BUN, Day 364: number analyzed (Participants) | 67 | 68 | 52 | 50
  BUN, Day 364: Unknown | 0 | 0 | 0 | 0
  BUN, Day 364: Below | 0 | 0 | 0 | 0
  BUN, Day 364: Within | 67 | 60 | 52 | 45
  BUN, Day 364: Above | 0 | 8 | 0 | 5

27. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination. This outcome included all the subjects who received 1 dose of the study product and the results were tabulated per age stratum.
Time Frame: Within 21 days after the first vaccination (Day 0 - Day 20)
Population: The analysis was performed on the Total Vaccinated cohort (TVc), which included all vaccinated subjects. The results were tabulated for the pooled groups and per age stratum, because until Day 21 no distinction was made in terms of study groups, since all subjects had received 1 dose of GSK2340272A vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 1D & 2D (18-60y) Sub-Group | GSK2340272A 1D & 2D (>60y) Sub-Group
Number analyzed (Participants) | 120 | 120
Participants
  Any AE(s) | 53 | 31
  Grade 3 AE(s) | 10 | 1
  Related AE(s) | 24 | 14

28. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination. The results were tabulated per age stratum.
Time Frame: Within 84 days after the first vaccination and 63 days after the second vaccination (Day 0 - Day 83)
Population: The analysis was performed on the Total Vaccinated cohort (TVc), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 68 | 70 | 52 | 50
Participants
  Any AE(s) | 45 | 46 | 39 | 30
  Grade 3 AE(s) | 13 | 9 | 10 | 7
  Related AE(s) | 15 | 10 | 9 | 7

29. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. The results were tabulated per age stratum.
Time Frame: During the entire study period (from Day 0 up to Day 364)
Population: The analysis was performed on the Total Vaccinated cohort (TVc), which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A 2D (18-60y) Sub-Group | GSK2340272A 2D (>60y) Sub-Group | GSK2340272A 1D (18-60y) Sub-Group | GSK2340272A 1D (>60y) Sub-Group
Number analyzed (Participants) | 68 | 70 | 52 | 50
Participants | 0 | 10 | 3 | 3

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: within the 84-day (Days 0-83) post-vaccination period; SAEs: during the entire study period (from Day 0 up to Day 364).
Arm/Group | GSK2340272A 1D Group | GSK2340272A 2D Group
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/138
Serious Adverse Events (participants affected / at risk) | 6/102 | 10/138
Other Adverse Events (participants affected / at risk) | 89/102 | 126/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2340272A 1D Group (N=102) | GSK2340272A 2D Group (N=138)
Aortic stenosis (Vascular disorders) | 0 | 1
Arrhytmia (Cardiac disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cervical root pain (Nervous system disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340272A 1D Group (N=102) | GSK2340272A 2D Group (N=138)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (16) | 35 (46)
Chills (General disorders) | 14 (14) | 29 (39)
Erythema (Skin and subcutaneous tissue disorders) | 8 (8) | 9 (11)
Fatigue (General disorders) | 30 (30) | 57 (77)
Headache (Nervous system disorders) | 35 (38) | 53 (75)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 (8) | 28 (33)
Myalgia (Musculoskeletal and connective tissue disorders) | 23 (23) | 48 (59)
Nasopharyngitis (Infections and infestations) | 20 (21) | 34 (39)
Pain (General disorders) | 80 (81) | 113 (196)
Swelling (General disorders) | 14 (14) | 14 (16)
Upper respiratory tract infection (Infections and infestations) | 7 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.